CLINICAL TRIAL: NCT03728296
Title: Clinical Study on the Safety and Efficacy of Autologous Induced Islet Body With Type 1 Diabetes
Brief Title: A Study of Autologous Induced Islet Body With Type 1 Diabetes
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: islet body-01
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- islet body treatment group (Experimental)
  Interventions: Biological: islet body

INTERVENTIONS:
Biological: islet body — Transplanting islet bodies under the diaphragm

SUMMARY:
This is a single centre、single arm、open-label study，to investigate the safety and efficacy of Autologous induced islet body With Type 1 diabetes

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years old (including 18 and 70 years old)
2. Diagnosed as type I diabetes, the diagnostic criteria refer to the 1990 WHO diabetes diagnostic criteria:

（1）Diabetes symptoms (hyperglycemia caused by polydipsia, polyphagia, weight loss, itchy skin, blurred vision and other acute metabolic disorders) + random blood glucose ≥ 11.1nmol / L; （2）Fasting blood glucose ≥7.0mmol/L or 75g glucose meets 2-hour blood glucose ≥11.1mmol/L.

3、Voluntary informed consent is given, agree to follow the trial treatment and visit plan.

Note: 2 is the venous plasma glucose level, if there is no diabetes symptoms, it is necessary to repeat the test on the next day.

Exclusion Criteria:

1. Patients with acute complications of diabetes: including diabetic ketosis, diabetic ketoacidosis, diabetes, hyperglycemia, hypertonic state, etc.
2. Patients with Severe bacterial and viral infections
3. patients are participating in other clinical trials and treating with other immune cellular products (DC, CIK, T, NK, and Car T products with CD19 or other targets)
4. Patients with severe cardiovascular and cerebrovascular disease (NYHA class 3-4) cannot cooperate with the study
5. Patients with severe liver dysfunction(liver function AST and ALT exceeded 2.5 times the normal upper limit).
6. Patients with kidney disease or moderate to severe renal insufficiency (renal function eGFR <60 ml/min/1.73 m2)
7. Women in pregnancy (urine/blood pregnancy test positive) or lactation; men or women with pregnancy plans in the last year; patients are not guaranteed to take effective contraceptive measures during the trial;
8. patients were diagnosed as tumor or tumor chemotherapy, radiotherapy and acute uric acid nephropathy within 5 years.
9. Other circumstances that researchers do not consider suitable for research.
10. Withdrawal from trial, loss of follow-up or death due to other reasons
11. Incomplete data, affecting effectiveness and safety judges
12. Researchers believe that the need for termination of the trial is needed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.0 | 1 year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment